CLINICAL TRIAL: NCT05627622
Title: Effectiveness of WhatsApp Education and Support Messages for Urolithiasis Prevention
Acronym: StoneApp
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Michael Frumer, Urology Resident, Principal Investigator, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: StoneApp
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Urinary Tract Stone
Keywords: Urinary Tract Stone; Kidney Stone; Health Education; Preventive Medicine
MeSH Terms: conditions — Urinary Calculi; Kidney Calculi; Health Education

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group, (Experimental): Receiving stone-prevention information on a monthly basis, using WhatsApp Messenger® application.
  Interventions: Behavioral: WhatsApp health education message
- control group (No Intervention): will not receive stone-prevention information

INTERVENTIONS:
Behavioral: WhatsApp health education message — stone-prevention information on a monthly basis, using personal WhatsApp messages
  Arms: Experimental group,

SUMMARY:
Kidney and ureteral stones are a common problem in primary care practice with increasing prevalence over the last few decades.

Prevention of recurrent stones (which are usually composed primarily of calcium oxalate) is aimed at decreasing the concentrations of the lithogenic factors. There are several metabolic and dietary treatable components. In all patients with urolithiasis, adequate fluid intake and lower body mass index are key components to reducing the risk of recurrent stones. For most patients, additional beneficial dietary modifications are increasing intake of fruits and vegetables which are rich in potassium, and reducing intake of candies and sweetened juices which are rich in sucrose and fructose. In addition, for patients who have been prescribed medications, adherence to medication may become an important issue over the long term.

Mobile technology has the potential to optimize health care and patient's adherence, especially through personal education and dissemination of health information. One of the most common technologies available on mobile is the WhatsApp Messenger® application. WhatsApp is a freeware messaging service; it allows streamlining patient-provider communication via text and voice messages, video clips and images.

The research hypotheses are, first, that use of WhatsApp to disseminate information regarding stones preventive measures will have a substantial positive effect on follow-up compliance and on patient's adherence to the preventive measures. Second, the investigators expect reduction in cumulative stone recurrence rate.

DETAILED DESCRIPTION:
Kidney and ureteral stones are a common problem in primary care practice with increasing prevalence over the last few decades. Nineteen percent of men and nine percent of women will be diagnosed with a kidney stone by the age of 70 years,and the rates of emergency department visit for urolithiasis were increased from 178 to 340 visits per 100,000 individuals from 1992 to 2009 (United States).

Prevention of recurrent stones, which are usually composed primarily of calcium oxalate, is aimed at decreasing the concentrations of the lithogenic factors. There are several metabolic and dietary treatable components. In all patients with urolithiasis, adequate fluid intake and lower body mass index are key components to reducing the risk of recurrent stones. For most patients, additional beneficial dietary modifications are increasing intake of fruits and vegetables which are rich in potassium, and reducing intake of candies and sweetened juices which are rich in sucrose and fructose. In addition, for patients who have been prescribed medications, adherence to medication may become an important issue over the long term.

As early as the 1980s, "The stone clinic effect" on the recurrence rate of stone disease was published. Hosking et al. demonstrated that a regimen of increased fluid intake and appropriate dietary modifications, to avoid dietary excesses, reduces stone growth and new stone formation in patients with idiopathic calcium urolithiasis.

According to the 2019 European Association of Urology guidelines on urolithiasis, all stone formers, independent of their individual risk, should follow preventive measures such as circadian fluid drinking of 2.5-3 liter daily, limitation of NaCl content to 5 gram daily.

The trials documenting benefit from these preventive measures required at least three years before the results were significant. However, in an analysis of over 3000 patients followed in a well-organized stone clinic at the University of Chicago, between 20% and 30% of patients were lost to follow-up every year. Only 15 to 40 percent of patients complied with the follow-up requirements by three years. Adherence to long-term therapy among those who did not follow-up was presumably very low. Hence, improving patient's adherence and follow-up compliance is of paramount importance.

Mobile technology has the potential to optimize health care and patient's adherence, especially through personal education and dissemination of health information. One of the most common technologies available on mobile is the WhatsApp Messenger® application. WhatsApp is a freeware messaging service; it allows streamlining patient-provider communication via text and voice messages, video clips and images.

The research hypotheses are, first, that use of WhatsApp to disseminate information regarding stones preventive measures will have a substantial positive effect on follow-up compliance and on patient's adherence to the preventive measures. Second, the investigators expect reduction in cumulative stone recurrence rate.

Methods Hypotheses will be tested in a randomized control trial. Participants will be recruited at the stone clinic of Rabin Medical Center, an academic tertiary hospital. Participants will randomly assign to one of two groups: A, the experimental group, receiving stone-prevention information on a monthly basis, and B, the control group.

Statistical Analysis Based on recurrence rates of previous studies the required number of patients was calculated in expectation of 20% and 40% cumulative recurrence rate of renal stones at 5 years in the experimental and control group, respectively. Type 1 error was set to 5%, and type 2 error was set to 20%. With this assumption, each group has to include 81 patients. Risk and rate ratio of stone recurrence and 95% confidence intervals (CIs) will be calculated. Loss of patients from follow-up will be measured by proportion of patients lost at each year.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to give informed consent
* Personal history of urolithiasis
* Stone free status
* A personal mobile phone with WhatsApp Messenger® application

Exclusion Criteria:

* Children
* Does not read Hebrew, the language in which the messages are written

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Stone recurrence | 5 years
  Rate of participants with urinary stone recurrence

SECONDARY OUTCOMES:
Mean time to relapse | 5 years
  Mean time to urinary stone event
Lost to follow-up rate | 5 years
  Rate of participants lost to follow-up in the urinary stone clinic

CONTACTS AND LOCATIONS:
Overall Officials: MIchael Frumer, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hosking DH, Erickson SB, Van den Berg CJ, Wilson DM, Smith LH. The stone clinic effect in patients with idiopathic calcium urolithiasis. J Urol. 1983 Dec;130(6):1115-8. doi: 10.1016/s0022-5347(17)51711-5. PMID 6644890
- [Background] Skolarikos A, Straub M, Knoll T, Sarica K, Seitz C, Petrik A, Turk C. Metabolic evaluation and recurrence prevention for urinary stone patients: EAU guidelines. Eur Urol. 2015 Apr;67(4):750-63. doi: 10.1016/j.eururo.2014.10.029. Epub 2014 Nov 20. PMID 25454613
- [Background] Ackermann D. Prophylaxis in idiopathic calcium urolithiasis. Urol Res. 1990;18 Suppl 1:S37-40. doi: 10.1007/BF00301526. PMID 2291248
- [Background] Sromicki J, Hess B. Simple dietary advice targeting five urinary parameters reduces urinary supersaturation in idiopathic calcium oxalate stone formers. Urolithiasis. 2020 Oct;48(5):425-433. doi: 10.1007/s00240-020-01194-7. Epub 2020 Jun 10. PMID 32524204